CLINICAL TRIAL: NCT06511934
Title: Intuitive, Complete Neural Control of Tablet Computers for Communication
Brief Title: Feasibility of the BrainGate2 Neural Interface System in Persons With Tetraplegia (BG-Tablet-01)
Acronym: BG-Tablet-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leigh R. Hochberg, MD, PhD. (Other)
Collaborators: Brown University (Other); Stanford University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Leigh R. Hochberg, MD, PhD., Neurologist, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2009P000505 (BG-Tablet-01); U01DC017844 (NIH)
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Brainstem Stroke; ALS; Tetraplegia; Spinal Cord Injuries; Cervical Spinal Cord Injury
MeSH Terms: conditions — Brain Stem Infarctions; Quadriplegia; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- BrainGate Neural Interface System (Experimental): Device: BrainGate Neural Interface System
  Interventions: Device: BrainGate Neural Interface System

INTERVENTIONS:
Device: BrainGate Neural Interface System — Placement of the BrainGate2 sensor(s) into arm-hand motor-related cortex.

SUMMARY:
People with brainstem stroke, advanced amyotrophic lateral sclerosis (ALS, also known as Lou Gehrig's disease), or other disorders can become unable to move or speak despite being awake and alert. In this project, the investigators seek to further translate knowledge about interpreting brain signals related to movement, and to further develop an intracortical brain-computer interface (iBCI) that could restore rapid and intuitive use of communication apps on tablet computers by people with paralysis.

DETAILED DESCRIPTION:
The goal of this project is to advance the methods by which people with tetraplegia can gain intuitive, reliable control of communication apps on industry-standard tablet computers through use of an intracortical brain-computer interface (iBCI).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of spinal cord injury, brainstem stroke, muscular dystrophy, amyotrophic lateral sclerosis or other motor neuron disorders
* Complete or incomplete tetraplegia (quadriplegia)
* Must live within a three-hour drive of the Study site
* Prior enrollment in BrainGate2 clinical trial (NCT00912041)

Exclusion Criteria:

* Visual impairment such that extended viewing of a computer monitor would be difficult even with ordinary corrective lenses
* Chronic oral or intravenous steroids or immunosuppressive therapy
* Other serious disease or disorder that could seriously affect ability to participate in the study

(There are additional exclusion criteria)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Sensor implant duration for at least one-year without any device-related Serious Adverse Events or explant | 1 year
  To determine the safety of the Sensor and overall safety of the System. Participants will be considered a success for this safety measure if they are successfully implanted with the Sensor(s) and:
  1. the sensors are not explanted for safety reasons during the one-year post-implant evaluation period.
  2. there are no device-related Serious Adverse Events that result in death or permanently increased disability during the one-year post-implant evaluation period.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh R Hochberg, MD, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Masssachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No